CLINICAL TRIAL: NCT03795376
Title: HIV Prevention in France : "Dat'AIDS Prevention"
Brief Title: Dat'Aids Prevention
Status: Recruiting | Type: Observational
Sponsor: DatAids (Other)
Responsible Party: Sponsor
Other Study IDs: DAT_002
Record Dates: First submitted 2018-12-21; First posted 2019-01-07 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: HIV Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
DatAIDS prevention is a cohort study of HIV prevention in over 23 HIV sites in France including overseas, aiming to describe HIV prevention in every aspect including HIV screening, STI and hepatitis screening, post-exposure prophylaxis and pre-exposure prophylaxis

ELIGIBILITY:
Inclusion Criteria:

* Male and female over 18 years old,
* HIV negative
* Attending for :
* HIV screening
* Hepatitis screening
* STI screening / treatment
* Blood, body fluid or sexual exposure
* Post-exposure prophylaxis
* Pre-exposure prophylaxis
* Signed consent

Exclusion Criteria:

* HIV-infection
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All persons attending for HIV prevention and seeking care at 23 centers using NADIS are included in the Dataids Prevention cohort after receiving oral information and giving written consent. NADIS is an electronic medical record (EMR) for HIV infection (and Hepatitis B virus (HBV), Hepatitis C virus (HCV), STI) and HIV prevention in French public hospitals.
  The Dataids Prevention study recruits persons HIV- and above the age of 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients enrolled for HIV prevention in the cohort | From date of enrollment, through study completion, an average of 1 year
  Demographics, risk factors clinical and biological characteristics, treatment of patients enrolled for HIV prevention in the cohort

SECONDARY OUTCOMES:
Proportion of persons enrolled for pre-exposure prophylaxis in the cohort | From date of enrollment, through study completion, an average of 1 year
  Demographics, risk factors clinical and biological characteristics, treatment of patients attending for pre-exposure prophylaxis in the cohort
Proportion of persons enrolled for post-exposure prophylaxis in the cohort | From date of enrollment, through study completion, an average of 1 year
  Demographics, risk factors clinical and biological characteristics, treatment of patients attending for post-exposure prophylaxis in the cohort
Proportion of persons enrolled for hepatitis screening in the cohort | From date of enrollment, through study completion, an average of 1 year
  Demographics, risk factors clinical and biological characteristics, treatment of patients attending for hepatitis screening in the cohort
Proportion of persons enrolled for pre-exposure prophylaxis in the cohort according to national French guidelines | From date of enrollment, through study completion, an average of 1 year
  Adequation between prevention practices and guidelines
Proportion of persons enrolled for post-exposure prophylaxis in the cohort according to national French guidelines | From date of enrollment, through study completion, an average of 1 year
  Adequation between prevention practices and guidelines
Incidence of STIs | From date of enrollment, through study completion, an average of 1 year
Incidence of hepatitis | From date of enrollment, through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pascal PUGLIESE, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice; André CABIE, MD-PhD, Principal Investigator — Centre Hospitalier Universitaire de Martinique
Locations (31):
- France (29):
  - Hôpital Nord Franche Comté, Belfort
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHRU Brest, Brest
  - CHU Clermont-Ferrand - Hôpital Gabriel-Montpied, Clermont-Ferrand
  - CHD Vendée, La Roche-sur-Yon
  - Hôpital Bicêtre - Assistance Publique des Hôpitaux de Paris, Le Kremlin-Bicêtre
  - CHU Limoges, Limoges
  - Hôpital de la Croix-Rousse - Hospices Civils de Lyon, Lyon
  - Hôpital Sainte Marguerite - Assistance Publique des Hôpitaux de Marseille, Marseille
  - IHU - Assistance Publique des Hôpitaux de Marseille, Marseille
  - CHR Metz-Thionville, Metz
  - Hôpital Gui de Chauliac, Montpellier
  - CHU Nancy - Hôpital Brabois, Nancy
  - CHU Nantes - Hôtel-Dieu, Nantes
  - CHU Nice - Hôpital l'Archet, Nice
  - CH Nîmes, Nîmes
  - CHR Orléans, Orléans
  - Groupe Hospitalier Pitié Salpêtrière - Assistance Publique des Hôpitaux de Paris, Paris
  - Hôpital Bichat - Assistance Publique des Hôpitaux de Paris, Paris
  - Hôpital Necker-Pasteur - Assistance Publique des Hôpitaux de Paris, Paris
  - Centre Hospitalier de Cornouaille, Quimper
  - CHU Reims - Hôpital Robert Debré, Reims
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU Rouen, Rouen
  - CHU St Etienne - Hôpital Nord, Saint-Etienne
  - CHU Strasbourg - Hôpital Civil, Strasbourg
  - CHU Toulouse - Hôpital Purpan, Toulouse
  - CHU Tourcoing - Hôpital Guy Chatiliez, Tourcoing
  - CH Bretagne-Atlantique, Vannes
- CHU de Guadeloupe, Pointe-à-Pitre, Guadeloupe
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No